CLINICAL TRIAL: NCT07112937
Title: The Effect of Multimodal Treatment of Rectal Cancer on Circulating Tumor Cells: A Prospective, Observational Study
Status: Recruiting | Type: Observational
Sponsor: The Institute of Molecular and Translational Medicine, Czech Republic (Other)
Responsible Party: Sponsor
Other Study IDs: 01/RVO-FNOs/2023; LF_2023_0118 (Other: Faculty of Medicine, Palacky University, Olomouc, Czechia)
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Rectal Cancer Patients
Keywords: circulating tumor cells
MeSH Terms: conditions — Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rectal cancer patients with neoadjuvant chemoradiotherapy
- Rectal cancer patients without neoadjuvant chemoradiotherapy

SUMMARY:
The prospective study will focus on patients undergoing multimodal treatment for rectal cancer. The main objective of the study will be to monitor changes in circulating tumor cells (CTCs) in the peripheral blood of patients during multimodal treatment. For each patient enrolled in the study, peripheral blood samples will be collected at specified time intervals to determine the presence and quantity of CTCs.

The CTCs levels will be compared among rectal cancer patients with neoadjuvant chemoradiotherapy and without neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria: rectal cancer -

Exclusion Criteria: no other cancer

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rectal cancer patients
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Levels of circulating tumor cells in peripheral blood | The levels of circulating tumor cells will be measured in 5 time points: before neoadjuvant chemoradiotherapy, in 3. week of chemoradioterapy, before surgery, one week after surgery and one month after surgery.
  The levels of circulating tumor cells will be measured in rectal cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ostrava, Ostrava, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Patients code; sex; age; diagnosis; clinical, laboratory and experimental findings
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Ihnat P, Srovnal J, Hrubovcak J, Martinek L. Detection and clinical significance of circulating tumour cells in patients with colorectal carcinoma. Rozhl Chir. 2023;102(10):376-380. doi: 10.33699/PIS.2023.102.10.376-380. PMID 38302423